CLINICAL TRIAL: NCT03876938
Title: Randomized, Placebo-controlled Trial of Olanzapine Versus Aprepitant Plus Ondansetron and Dexamethasone as Antiemetic Prophylaxis in Patients Receiving High Emetic Chemotherapy
Brief Title: Olanzapine Versus Aprepitant Based Antiemetic Regimen for High Emetic Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 728/2561(EC4)
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Antiemetic for Highly Emetogenic Chemotherapy
MeSH Terms: interventions — Aprepitant; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aprepitant (Active Comparator): aprepitant / dexamethasone/ ondansetron
  Interventions: Drug: aprepitant
- olanzapine 10 mg (Experimental): olanzapine 10 mg/dexamethasone/ ondansetron
  Interventions: Drug: olanzapine 10 mg
- olanzapine 5 mg (Experimental): olanzapine 5 mg/dexamethasone/ ondansetron
  Interventions: Drug: olanzapine 5 mg

INTERVENTIONS:
Drug: aprepitant — aprepitant 125 mg orally, dexamethasone 12 mg iv, ondansetron 8 mg iv before chemotherapy aprepitant 80 mg orally D2-4, dexamethasone 8 mg/day orally D2-4
  Arms: aprepitant
Drug: olanzapine 10 mg — olanzapine 10 mg orally, dexamethasone 12 mg iv, ondansetron 8 mg iv before chemotherapy olanzapine 10 mg orally D2-4, dexamethasone 8 mg/day orally D2-4
  Arms: olanzapine 10 mg
Drug: olanzapine 5 mg — olanzapine 5 mg orally, dexamethasone 12 mg iv, ondansetron 8 mg iv before chemotherapy olanzapine 5 mg orally D2-4, dexamethasone 8 mg/day orally D2-4
  Arms: olanzapine 5 mg

SUMMARY:
Aprepitant and olanzapine have been recommended for emesis prevention from highly emetogenic chemotherapy. We hypothesized that olanzapine may lead to less nausea compared to aprepitant based on previous study. However, data of combination of olanzapine and ondansetron is scarce.

DETAILED DESCRIPTION:
Aprepitant and olanzapine have been recommended for emesis prevention from highly emetogenic chemotherapy. We hypothesized that olanzapine may lead to less nausea compared to aprepitant based on previous study. However, data on efficacy and adverse effects of combination of olanzapine and ondansetron which is only serotonin antagonist in Thai national essential drug list, is scarce. Also, we aims to assess the efficacy of olanzapine dosage of 5 mg which is more commonly used in Thai patients.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proved of solid malignancy
* receive first cycle of cisplatin >= 50 mg/m2 or cyclophosphamide/doxorubicin

Exclusion Criteria:

* pregnancy
* patients with episode of vomiting within 24 hours before starting chemotherapy
* uncontrolled brain/ CNS metastasis
* gut obstruction
* receive combination of moderate or high emetogenic chemotherapy during Day 2-5
* Known allergy to ondansetron, olanzapine, aprepitant or dexamethasone
* currently receive olanzapine with other indication and plan to continue the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
no nausea rate | Days 1-5 of chemotherapy
  proportion of patients report no nausea

SECONDARY OUTCOMES:
complete remission | Days 1-5 of chemotherapy
  no episode of vomiting
>= grade 3 vomiting | Days 1-5 of chemotherapy
  higher than grade 3 vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Suthinee Ithimakin, MD, Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Division of medical oncology, department of medicine Siriraj Hospital, Bangkok
  - Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No